CLINICAL TRIAL: NCT01963143
Title: A Phase III, Multicenter, Open-label, Randomized, Two-Period, Crossover Bioequivalence Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Gammaplex® 10 and Gammaplex® 5% in Primary Immunodeficiency Diseases
Brief Title: Bioequivalence Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Gammaplex® 10 and Gammaplex® 5% in Primary Immunodeficiency Diseases
Acronym: GMX07
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio Products Laboratory (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GMX07
Record Dates: First submitted 2013-09-13; First posted 2013-10-16 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Primary Immune Deficiency Disorders; Common Variable Immunodeficiency; X-linked Agammaglobulinaemia; Hyper-IgM Syndrome
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Common Variable Immunodeficiency; Bruton type agammaglobulinemia; Hyper-IgM Immunodeficiency Syndrome | interventions — gamma-Globulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Sequence 1 - Adults (Experimental): Gammaplex 5% - 5 intravenous infusions at a dose of 300 to 800 mg/kg/infusion, given every 21 to 28 days, followed by Gammaplex 10 - 5 intravenous infusions at a dose of 300 to 800 mg/kg/infusion, given every 21 to 28 days
  Interventions: Biological: Gammaplex (5%); Biological: Gammaplex 10
- Treatment Sequence 2 - Adults (Experimental): Gammaplex 10 - 5 intravenous infusions at a dose of 300 to 800 mg/kg/infusion, given every 21 to 28 days, followed by Gammaplex 5% - 5 intravenous infusions at a dose of 300 to 800 mg/kg/infusion, given every 21 to 28 days
  Interventions: Biological: Gammaplex (5%); Biological: Gammaplex 10
- Pediatrics (Experimental): Gammaplex 10 - 5 intravenous infusions at a dose of 300 to 800 mg/kg/infusion, given every 21 to 28 days
  Interventions: Biological: Gammaplex 10

INTERVENTIONS:
Biological: Gammaplex (5%)
  Arms: Treatment Sequence 1 - Adults; Treatment Sequence 2 - Adults
Biological: Gammaplex 10

SUMMARY:
The primary objective is to demonstrate the bioequivalence of Gammaplex® 10 intravenous immunoglobulin (IGIV) and Gammaplex® 5% IGIV with respect to area under the curve within a 28-day dosing interval (AUC0-28) in a cohort of adult subjects.

The secondary objectives are to demonstrate the bioequivalence of Gammaplex® 10 IGIV and Gammaplex® 5% IGIV with respect to area under the curve within a 21-day dosing interval (AUC0-21) in adult subjects; to assess the pharmacokinetics of Gammaplex 10 IGIV and Gammaplex 5% IGIV including Immunoglobulin G (IgG) trough levels and to investigate the safety and tolerability of Gammaplex 10 IGIV and Gammaplex 5% IGIV in adults subjects; to assess the pharmacokinetics of Gammaplex 10 IGIV including IgG trough levels and to investigate the safety and tolerability of Gammaplex 10 IGIV in pediatric subjects.

ELIGIBILITY:
Inclusion criteria:

1. Adult cohort: The subject is aged 16 to 55 years inclusive, is of either sex, and belongs to any ethnic group.

   Pediatric cohort: The subject is aged 2 to 15 years inclusive, is of either sex, weighs at least 10 kg, and belongs to any ethnic group.
2. The subject has primary immunodeficiency disease, e.g. common variable immunodeficiency, X linked and autosomal forms of agammaglobulinemia, hyper IgM (Immunoglobulin M) syndrome. Isolated deficiency of a single IgG subclass or of specific antibodies without hypogammaglobulinemia per se, does not qualify for inclusion.
3. The subject is currently receiving a licensed IGIV (or investigational stage III, IIIb IGIV) at a dose that has not changed by ± 50% of the mean dose for at least three months before study entry and is between 300 and 800 mg/kg/infusion. The infusion interval must be either every 21 or every 28 days.
4. The subject must have a trough level ≥ 6 g/L (600 mg/dL). At least one documented trough level must be available from the three months before Screening.
5. The subject must have documentation from the last three consecutive routine IGIV infusions for the following, before the first infusion in this study: dose of IGIV, treatment intervals, and trade name (or identity) of the IGIV treatment.
6. Female subjects of childbearing potential must have a negative result on an HCG (human chorionic gonadotropin) based pregnancy test at Screening.
7. Females who are or become sexually active must practice contraception using a method of proven reliability for the study duration.
8. The subject is willing to comply with all aspects of the protocol for the duration of the study.
9. The subject has signed an informed consent form and assent form (if applicable).

Exclusion criteria:

1. The subject has a history of any severe anaphylactic reaction to blood or any blood derived product.
2. The subject has selective IgA deficiency, history of reaction to products containing IgA (Immunoglobulin A), or has a history of antibodies to IgA.
3. The subject has cellular or innate impaired immunity (i.e. only subjects with humoral impaired immunity may be included).
4. The subject has evidence of an active infection at the time of enrolment.
5. The subject has previously completed or withdrawn from this study.
6. The subject is currently receiving, or has received, any investigational agent other than an IGIV within the prior three months.
7. The subject is pregnant or is nursing.
8. The subject has positive results for any of the following at Screening:

   * Serological test for HIV 1 and 2, HCV, or HBsAg
   * NAT (Nucleic acid amplification technique)for HCV
   * NAT for HIV
9. The subject has levels > 2.5 times the upper limit of normal, as defined at the central laboratory, of any of the following at Screening:

   * Alanine amino transaminase
   * Aspartate amino transaminase
10. The subject has severe renal impairment (defined as serum creatinine greater than two times the upper limit of normal or blood urea nitrogen greater than 2.5 times the upper limit of normal for the range of the laboratory doing the analysis); the subject is on dialysis; the subject has a history of acute renal failure.
11. The subject is known to abuse alcohol, opiates, psychotropic agents, or other chemicals or drugs, or has done so within the past 12 months.
12. The subject has a history of deep vein thrombosis or thrombotic complications of IGIV therapy.
13. The subject suffers from any acute or chronic* medical condition (e.g. renal disease or predisposing conditions for renal disease, coronary artery disease, or protein losing state) that the Investigator feels may interfere with the conduct of the study.
14. The subject has an acquired immunodeficiency condition such as chronic* lymphocytic leukemia, lymphoma, multiple myeloma, or chronic or recurrent neutropenia (absolute neutrophil count < 1 × 109/L).
15. The subject is receiving the following medication:

    * Steroids (long term daily, ≥ 0.15 mg of prednisone equivalent/kg/day). Requirement for short or intermittent courses of steroids would not exclude a subject.
    * Immunosuppressive drugs
    * Immunomodulatory drugs
16. The subject has uncontrolled arterial hypertension (systolic blood pressure > 160 mm Hg and/or diastolic blood pressure > 100 mm Hg).
17. The subject has anemia (hemoglobin < 10 g/dL) at Screening.
18. The subject is known to be intolerant to any component of Gammaplex, such as sorbitol (i.e. hereditary intolerance to fructose) or glycine.

    * Chronic conditions would be as per the Investigator's opinion however for this study the guidance is that the condition has been present for at least 6 months.

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wolford, Study Director — Bio Products Laboratory
Locations (17):
- United States (14):
  - Arizona Allergy Associates, Chandler, Arizona
  - Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Allergy Associates of the Palm Beaches, PA, North Palm Beach, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Institute for Asthma and Allergy, Chevy Chase, Maryland
  - Asthma and Allergy Center, Toledo, Ohio
  - Dallas Allergy Immunology Research, Dallas, Texas
  - University of Utah Primary Children's Hospital, Salt Lake City, Utah
  - O&O Alpan, LLC, Fairfax, Virginia
  - Bellingham Asthma Allergy and Immunology Clinic, Bellingham, Washington
- Egyesitett Szent Istvan es Szent Laszlo Korhaz, Budapest, Hungary
- United Kingdom (2):
  - University Hospital of Wales, Cardiff, Wales
  - The Royal Free Hospital and Medical School, London

REFERENCES:
- [Derived] Rajendram V, Paddick M, More J. Measles neutralising antibody levels in patients receiving intravenous immunoglobulin treatment - a sub-analysis of a randomized, cross-over bioequivalence trial. PLoS One. 2025 Feb 7;20(2):e0316926. doi: 10.1371/journal.pone.0316926. eCollection 2025. PMID 39919133
- [Derived] Geng B, Clark K, Evangelista M, Wolford E. Low rates of headache and migraine associated with intravenous immunoglobulin infusion using a 15-minute rate escalation protocol in 123 patients with primary immunodeficiency. Front Immunol. 2023 Feb 2;13:1075527. doi: 10.3389/fimmu.2022.1075527. eCollection 2022. PMID 36818468

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence 1 - Adults: Gammaplex 5% & Gammaplex 10 on a 21-day treatment schedule
- Treatment Sequence 2 - Adults: Gammaplex 10 and Gammaplex 5% on a 28-day treatment schedule
- Pediatrics: Gammaplex 10 on a 21 or 28 day treatment schedule
Period: Overall Study
Arm/Group | Treatment Sequence 1 - Adults | Treatment Sequence 2 - Adults | Pediatrics
Started | 14 | 19 | 15
Completed | 14 | 18 | 14
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Sequence 1 - Adults: Gammaplex 5% and Gammaplex 10 on a 21-day schedule
- Treatment Sequence 2 - Adults: Gammaplex 5% and Gammaplex 10 on a 28-day schedule
- Pediatrics: Gammaplex 10 on a 21 or 28 day schedule
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 - Adults | Treatment Sequence 2 - Adults | Pediatrics | Total
Number analyzed (Participants) | 14 | 19 | 15 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 15 | 17
  Between 18 and 65 years | 13 | 18 | 0 | 31
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 7 | 28
  Male | 2 | 10 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 14 | 18 | 13 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 14 | 19 | 15 | 48
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 0 | 0 | 1 | 1
  United States | 11 | 19 | 14 | 44
  United Kingdom | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Primary Bioequivalence Analysis - Area Under the Curve Within a 28-day Dosing Interval (AUC0-28) in Adult Subjects
Time Frame: After a minimum 5 infusions on each product, at pre-infusion, 10 minutes before end of infusion, 1, 3, 6, 24, 48 hours, 4, 7, 14, 21 and 28 days post-infusion
Population: PK population
Measure: Geometric Mean (90% Confidence Interval); unit: ratio Gammaplex 10%/Gammaplex 5%
Arm/Group | Gammaplex 10% | Gammaplex 5%
Number analyzed (Participants) | 16 | 16
ratio Gammaplex 10%/Gammaplex 5%
  AUC(0-t) absolute | 1.01 [0.98 to 1.03] | 1.01 [0.98 to 1.03]
  AUC(0-t) baseline-adjusted | 1.07 [0.93 to 1.23] | 1.07 [0.93 to 1.23]

2. Secondary Outcome: Secondary Bioequivalence Analysis - Area Under the Curve Within a 21-Day Dosing Interval (AUC0-21) in Adult Subjects
Time Frame: After a minimum 5 infusions on each product, at pre-infusion, 10 minutes before end of infusion, 1, 3, 6, 24, 48 hours, 4, 7, 14 and 21 days post-infusion
Measure: Geometric Mean (90% Confidence Interval); unit: ratio Gammaplex 10%/Gammaplex 5%
Arm/Group | Gammaplex 10% | Gammaplex 5%
Number analyzed (Participants) | 14 | 14
ratio Gammaplex 10%/Gammaplex 5%
  AUC(0-t) absolute | 0.99 [0.95 to 1.02] | 0.99 [0.95 to 1.02]
  AUC(0-t) baseline-adjusted | 1.10 [0.96 to 1.26] | 1.10 [0.96 to 1.26]

3. Secondary Outcome: Secondary Bioequivalence Analysis - IgG Trough Levels
Time Frame: After a minimum 5 infusions on each product, at pre-infusion.
Measure: Geometric Mean (90% Confidence Interval); unit: ratio Gammaplex 10%/Gammaplex 5%
Arm/Group | Gammaplex 10% | Gammaplex 5%
Number analyzed (Participants) | 30 | 30
ratio Gammaplex 10%/Gammaplex 5%
  28-day dosing interval | 0.98 [0.94 to 1.02] | 0.98 [0.94 to 1.02]
  21-day dosing interval | 0.95 [0.92 to 0.99] | 0.95 [0.92 to 0.99]

ADVERSE EVENTS:
Groups:
- Gammaplex 5% - All Subjects: Subjects aged 17-55 years
- Gammaplex 10% - All Subjects: Subjects aged 2-55 years
Arm/Group | Gammaplex 5% - All Subjects | Gammaplex 10% - All Subjects
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/47
Serious Adverse Events (participants affected / at risk) | 2/33 | 1/47
Other Adverse Events (participants affected / at risk) | 23/33 | 44/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gammaplex 5% - All Subjects (N=33) | Gammaplex 10% - All Subjects (N=47)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gammaplex 5% - All Subjects (N=33) | Gammaplex 10% - All Subjects (N=47)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 8 (8)
Nasopharyngitis (Infections and infestations) | 1 (2) | 5 (7)
Viral upper respiratory tract infection (Infections and infestations) | 4 (5) | 4 (5)
Acute sinusitis (Infections and infestations) | 5 (6) | 3 (3)
Chronic sinusitis (Infections and infestations) | 2 (2) | 4 (4)
Sinusitis (Infections and infestations) | 1 (1) | 7 (7)
Influenza (Infections and infestations) | 0 (0) | 6 (6)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 6 (16) | 11 (28)
Migraine (Nervous system disorders) | 3 (4) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 3 (7) | 1 (5)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days